CLINICAL TRIAL: NCT02662283
Title: Validity and Security of Reh-acteoside Therapy for Patients of IgA Nephropathy -- A Prospective, Randomized, Controlled, Multi-Center Clinical Trial
Brief Title: Validity and Security of Reh-acteoside Therapy for Patients of IgA Nephropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, The Sixth Affiliated Hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usix-IgAN-002
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: IGA Nephropathy
Keywords: IGA Nephropathy; proteinurien; Reh-acteoside; Prednisolone
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prednisolone (Active Comparator): Oral take prednisolone (0.5 mg/kg, qd) for 8 weeks
  Interventions: Drug: Prednisolone
- Reh-acteoside (Experimental): Oral take reh-acteoside (0.4g bid) for 8 weeks
  Interventions: Drug: Reh-acteoside
- Reh-acteoside+Prednisolone (Experimental): Oral take prednisolone (0.5 mg/kg, qd) and reh-acteoside (0.4g bid) for 8 weeks
  Interventions: Drug: Prednisolone; Drug: Reh-acteoside

INTERVENTIONS:
Drug: Prednisolone — Oral take prednisolone (0.5 mg/kg, qd) for 8 weeks
  Arms: Prednisolone; Reh-acteoside+Prednisolone
Drug: Reh-acteoside — Oral take and reh-acteoside (0.4g bid) for 8 weeks
  Arms: Reh-acteoside; Reh-acteoside+Prednisolone

SUMMARY:
This prospective, randomized, controlled, multi-center clinical trial will evaluate the effect and security of reh-acteoside therapy for patients of IgA nephropathy.

DETAILED DESCRIPTION:
Reh-acteoside (general acteoside of rehmanniae leaves) contains more than 10 kinds of bio-active mucopolysaeccharide, among which acteoside is the most effective ingredient, constituting 30 percent. It has been reported that acteoside can reduce mesangium lesion of IgA nephrology-model ddy-mice, mainly by reducing the expressing of TGF-β1, reducing proliferation of mesangial cell and glomerular sclerosis. Research also suggested that conjunctive use of reh-acteoside and benazepril showed better effect on reducing proteinurine than single use of benazepril, with no obvious side effect at the same time. Thus, we start this clinical trial to evaluate the effect and security of reh-acteoside therapy for patients of IgA nephropathy. We set 3 groups: methylprednisolone group, reh-acteoside group and methylprednisolone with reh-acteoside group. After followed-up for 8 weeks, remission of proteinuria and change of renal function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Age 14~70 years, regardless of gender Clinical evaluation and renal biopsy diagnostic for IgA nephropathy. Average urinary protein excretion of 1.0~3.5g/24h on two successive examinations.

eGFR ≥ 50 ml/min/1.73 m2 Willingness to sign an informed consent (patients under 18 years old need legal guardian to sign).

Exclusion Criteria:

Secondary IgAN such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B -associated nephritis.

Rapidly progressive nephritic syndrome (crescent formation≥50%). Acute renal failure, including rapidly progressive IgAN. Renal biopsy suggests active pathological change (cellular crescent, loop necrosis, micro-thrombosis formation) Current or recent (within 30 days) exposure to steroids or immunosuppressive therapy (CTX、MMF、CsA、FK506).

Recent acute hepatitis (in 2 weeks), chronic active hepatitis (hepatitis B or hepatitis C infection), a rise more than 2.5 folds of current ALT, AST or TBil level.

History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease).

Any Active systemic infection or history of serious infection within one month. Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure , chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases).

Active tuberculosis Malignant hypertension that is difficult to be controlled by oral drugs. Known allergy, contraindication or intolerance to the steroids. Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception.

Malignant tumors Excessive drinking or drug abuse Mental aberrations Current or recent (within 30 days) exposure to any other investigational drugs.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Remission of proteinuria (complete or partial) | up to 8 weeks
  Complete remission: UPCR (urinary protein creatinine ratio) <300mg/g, plasma albumin in normal range, and stable serum creatinine level (fluctuation range <15%)； Partial remission: UPCR decreases more than 50% from baseline, plasma albumin >30g/L, and stable serum creatinine level (fluctuation range <15%).

SECONDARY OUTCOMES:
Deterioration of renal function | up to 8 weeks
  evidenced by a 50% rise from baseline serum creatinine (SCr) levels, or a 25% decline from baseline eGFR levels, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation
Deacrase of hematuria | up to 8 weeks
  urine RBC decreases more than 50% from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zongpei Jiang, M.D. & Ph.D., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Nephrology, 6th Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639